CLINICAL TRIAL: NCT06268080
Title: Preserving Brain Health After Surgery: Does Light General Anesthesia Reduce Postoperative Delirium and Cognitive Decline Compared With Deep General Anesthesia in Older Adults?
Brief Title: Depth of Anesthesia on Postoperative Delirium and Cognitive After Surgery
Acronym: Balanced-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auckland City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: A+9317
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Delirium, Postoperative; Anesthesia; Surgery-Complications; Cognition Disorder; Delirium; Cognitive Decline
Keywords: randomized controlled trial; multicentre; clinical trial; depth of anaesthesia; postoperative delirium
MeSH Terms: conditions — Emergence Delirium; Cognition Disorders; Delirium; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Multicentre, prospective, randomized, active control, parallel group, intention to treat, safety and efficacy study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding of procedural anesthesiologist is not possible. Patients, surgeons, and all outcome assessors will be blinded. One unblinded research coordinator at each site will collect pEEG related data points. Other research coordinators will be blinded as to treatment allocation and will collect data relating to primary and secondary outcomes. Clinicians carrying out participant usual care will be able to unblind study allocation if necessary by viewing the patients anesthesia record via password protected, accessing clinician identity logged, Electronic Health Record (EHR). This record will be unavailable for access by other means.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Light general anesthesia (Experimental): Bispectral Index (BIS) of 55
  Interventions: Behavioral: Depth of anesthesia titration using pEEG
- Deep general anesthesia (Active Comparator): Bispectral Index (BIS) of 40
  Interventions: Behavioral: Depth of anesthesia titration using pEEG

INTERVENTIONS:
Behavioral: Depth of anesthesia titration using pEEG — Titration of maintenance anesthetic agent (propofol infusion)

SUMMARY:
The goal of this clinical trial (Balanced-2 study) is to compare light to deep general anesthesia using widely available brain monitors, to see if 'light' anesthesia could reduce rates of delirium, cognitive decline, and disability in older adults undergoing major surgery.

Delirium is the most common serious surgical complication, occurring in an estimated one in four older adults undergoing major surgery. Delirium causes significant distress to patients and family, and is associated with prolonged hospital stay, physical disability, progression to dementia-like illnesses, and discharge to long-term care. Between 10 - 30% of adults aged 70 years and above have surgery every year, and preserving brain health and wellbeing is an important priority during this time.

Older adults (aged ≥65 years, or Indigenous, Pacific patients aged ≥55 years) undergoing major surgery with general anesthesia (excluding heart and brain surgery) and able to provide consent will be able to participate. Participants will be randomized to two groups - a lighter general anesthesia group and a deeper general anesthesia group using processed electroencephalography (a brain monitor that provides information on depth of anesthesia using brain waves). The anesthesiologist will titrate anesthetic drugs according to the brain monitor. Participants will be followed up to determine if they experience delirium after surgery, and longer term impact of delirium such as cognitive and physical decline will also be measured.

If found to be effect, this simple, cheap, and widely available treatment could reduce disability, preserve brain health and wellbeing of many older adults undergoing surgery worldwide, and save millions in healthcare dollars.

DETAILED DESCRIPTION:
The Balanced-2 study is a randomized clinical trial studying the effects of depth of anesthesia on the incidence of postoperative delirium, and its associated longer-term impact including cognitive, physical decline and mortality. The study follows accumulating evidence that titrating general anesthesia (GA) using processed electroencephalography (pEEG) can reduce the incidence of postoperative delirium, and has the most immediate promise as a preventative strategy.

The evidence to date is limited by 1) significant statistical heterogeneity between studies, 2) poor adherence to the intervention, resulting in poor or no separation between the intervention and standard care groups in some studies, 3) exclusion of high risk patients such as those with cognitive impairment, 4) evidence limited to inhalation anesthetic agents only.

The Balanced-2 study will recruit participants who are at higher risk of postoperative delirium (based on eligibility criteria), undergoing major surgery with total intravenous anesthesia (TIVA), with robust processes to ensure adherence and group separation. Participants will be randomized in a 1:1 ratio using a web-based service in permuted blocks of 8 patients according to region and stratified by surgical urgency and pre-existing neurocognitive disorders, to either light GA or deep GA from 10 mins after induction of anesthesia to emergence. Depth of anesthesia will be titrated using pEEG monitors such as the commonly used Bispectral index (BIS) and Patient State Index (PSI). The procedural anesthesiologist will pre-specify an individual mean arterial pressure (MAP) target before randomisation to avoid confounding. There will be limitations on the use of ketamine, nitrous oxide, clonidine and dexmedetomidine due to interference with pEEG, but all other aspects of care are determined by the procedural anesthesiologist or according to standard institutional protocol.

The sample size was based on calculations using the minimum clinically important effect size, as determined by a Delphi process with 2 stakeholder groups. A statistical analysis plan will be published prior to trial commencement.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 65 years, and Māori, Pacific or Indigenous participants aged ≥ 55 years who are undergoing major elective or non-elective surgery with expected surgical duration ≥ 2 hours and postoperative hospital stay ≥ 2 nights.
* Having general anesthesia using total intravenous anesthesia (TIVA) with pEEG monitoring
* Able to provide informed consent (including patients with mild preoperative neurocognitive disorders)

Exclusion Criteria:

* Intracranial or cardiac surgery
* Undergoing surgery with 'wake up' test
* Previous enrollment in Balanced-2 study
* Terminal illness with expected survival <3 months
* Emergency surgery within 6 hours of presentation to hospital
* Cognitive impairment with no capacity to consent or activated enduring power of attorney
* Clinically impaired and unable to consent due to acute pathology or preoperative delirium

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2766 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium (POD) | Administered twice a daily for up to 3 postoperative days or until discharge if discharge occurs before day 3, including weekends. Further once daily testing from days 4 to 7 if screens positive.
  Assessed using the Three-minute Diagnostic Interview for the Confusion Assessment Method (3D-CAM) or if patients are in the intensive care unit (ICU), the Confusion Assessment Method for the ICU (CAM-ICU). Delirium testing will occur between 0600 and 1000 and 1800 to 2200 daily including weekends.
  Delirium is present if both features (1) altered mental status/fluctuating course and (2) inattention are present, and features (3) altered level of consciousness, OR (4) disorganized thinking are present.

SECONDARY OUTCOMES:
Incidence of severe delirium | 7 days after surgery
  Assessed using Confusion Assessment Method - Severity Short Form (CAM-S)
  The CAM-S uses the 4 features of delirium and rates them as absent, mild or marked. Possible scores are o to 7, with higher scores indicating more severe delirium.
Incidence of new mild and major postoperative neurocognitive disorders | Assessed at 90 days and 1 year after surgery
  Diagnosis of new postoperative neurocognitive disorder requires 1) subjective complaint using standardized questionnaire, 2) objective testing using Mini-Addenbrooke's Cognitive Examination (ACE), and for a diagnosis of major postoperative neurocognitive disorder, 3) evidence of functional decline using Lawton-Brody's instrumental activities of daily living (ADL) scale.
  The Mini-ACE questionnaire is scored out of 30, with lower scores indicating more severe cognitive impairment. The Lawton-Brody's instrumental ADL scale is scored out of 8 for women, and 5 for men, with higher scores indicating more independence.
Postoperative cognitive decline | Assessed at 90 days and 1 year after surgery
  Defined by a 2 or more-point drop in Mini-Addenbrooke's Cognitive Examination scores.
  The Mini-ACE questionnaire is scored out of 30, with lower scores indicating more severe cognitive impairment.
Functional decline | Assessed at 90 days and 1 year after surgery
  As measured by the change in Lawton-Brody's instrumental ADL scores
  The Lawton-Brody's instrumental ADL scale is scored out of 8 for women, and 5 for men, with higher scores indicating more independence.
All-cause mortality | Assessed at 1 year after surgery
Duration of delirium | 7 days after surgery
  Duration of delirium for the first 7 days after surgery

OTHER OUTCOMES:
Incidence of awareness | Assessed once, between postoperative days 1 to 3
  Assessed using Brice questionnaire.
  The Brice questionnaire uses 6 questions to determine if there was risk of awareness under general anesthesia.
Adverse and serious adverse events | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Deng, Principal Investigator — Auckland City Hospital, Health New Zealand
Locations (3):
- New Zealand (3):
  - Auckland City Hospital, Health New Zealand, Grafton, Auckland
  - North Shore Hospital, Auckland, North Island
  - Christchurch Hospital, Christchurch, South Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evered LA, Chan MTV, Han R, Chu MHM, Cheng BP, Scott DA, Pryor KO, Sessler DI, Veselis R, Frampton C, Sumner M, Ayeni A, Myles PS, Campbell D, Leslie K, Short TG. Anaesthetic depth and delirium after major surgery: a randomised clinical trial. Br J Anaesth. 2021 Nov;127(5):704-712. doi: 10.1016/j.bja.2021.07.021. Epub 2021 Aug 28. PMID 34465469
- [Background] Sumner M, Deng C, Evered L, Frampton C, Leslie K, Short T, Campbell D. Processed electroencephalography-guided general anaesthesia to reduce postoperative delirium: a systematic review and meta-analysis. Br J Anaesth. 2023 Feb;130(2):e243-e253. doi: 10.1016/j.bja.2022.01.006. Epub 2022 Feb 17. PMID 35183345
- [Background] Deng C, Sidebotham D. Using the Delphi process to determine the minimum clinically important effect size for the Balanced-2 randomised controlled trial. Clin Trials. 2023 Oct;20(5):473-478. doi: 10.1177/17407745231173058. Epub 2023 May 5. PMID 37144615
- [Background] Evered L, Silbert B, Knopman DS, Scott DA, DeKosky ST, Rasmussen LS, Oh ES, Crosby G, Berger M, Eckenhoff RG; Nomenclature Consensus Working Group. Recommendations for the nomenclature of cognitive change associated with anaesthesia and surgery-2018. Br J Anaesth. 2018 Nov;121(5):1005-1012. doi: 10.1016/j.bja.2017.11.087. Epub 2018 Jun 15. PMID 30336844